CLINICAL TRIAL: NCT02775071
Title: Psychopathology, Disordered Eating, and Impulsivity as Predictors of Outcomes of Bariatric Surgery
Acronym: SIDE-BAR
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Kelly Allison, Associate Professor, University of Pennsylvania
Other Study IDs: 823735
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will evaluate the relationship between psychopathology, disordered eating, and impulsivity (measured by clinical interview, self-report measures, and objective testing) on changes in weight and psychosocial status in the first two years after bariatric surgery. Participants will be 300 adults who plan to undergo bariatric surgery. Participants will complete four assessments over a two-year period, one at baseline (before surgery) and 6, 12, and 24 months after surgery. Each assessment will include computer tasks, surveys, clinical interview, urine test, waist circumference and height/weight measurement. The investigators will track how psychopathology, disordered eating, and impulsivity are related to changes in weight and psychosocial status following bariatric surgery.

DETAILED DESCRIPTION:
Psychosocial Status and Psychopathology in Candidates for Bariatric Surgery:

Extreme obesity is associated with a signiﬁcant psychosocial burden, including impairments in quality of life, body image, sexual behavior and other areas of psychosocial functioning. While this distress is believed to contribute to the decision to have bariatric surgery, its impact on postoperative outcomes is less clear. At present, little is known about the physiological and behavioral contributions to success or failure of bariatric surgery. Regardless, weight regain after bariatric surgery is frequently attributed to preoperative psychosocial and behavioral factors. More speciﬁcally, there has been a great deal of interest in the presence of formal psychopathology in bariatric surgery patients and its potential contribution to postoperative outcomes. At least six studies have described rates of psychopathology in candidates for bariatric surgery using structured diagnostic instruments. Lifetime rates of any psychiatric diagnoses ranged from 36.8%-72.6%, higher than those reported in most studies of the general population. Mood disorders were the most frequent diagnoses, seen in 22.0%-54.8% of patients. Substance use disorders (SUDs) were found in up to 35.7% of patients and alcohol abuse or dependence in up to 33.2%. Binge eating disorder (BED), deﬁned as eating an unusually large amount of food within a short period of time coupled with a loss of control over eating, has been diagnosed in 4.6% to 27.1% of patients. Current diagnoses (as compared with lifetime) were less common, reported in 20.9%-55.5% of candidates for surgery. Mood disorders were diagnosed in up to 31.5%. BED ranged from 3.4%-41.9%. Current substance use was seen in less than 2% of patients. (Note. The lower percentages of those with current psychopathology, as opposed to lifetime psychopathology, are expected.) While studies of the psychosocial characteristics of bariatric surgery candidates have been informative, they are not without limitations. Many studies have suffered from methodological concerns, including small sample sizes or lack of an appropriate comparison group. Further, establishing psychiatric diagnoses prior to bariatric surgery is challenging. Perioperative guidelines suggest that patients undergo an evaluation with a mental health professional prior to surgery and most third party payers require these evaluations. However, most programs do not use structured clinical interviews to establish diagnoses for clinical purposes. Several studies have suggested that candidates for bariatric surgery engage in impression management prior to surgery, in which they minimize reports of psychopathology to present themselves to the bariatric team in the most favorable light. To address this issue, assessment of psychiatric symptoms for research purposes is recommended to occur independently from the required clinical evaluation, as the investigators will do in the proposed study. Nevertheless, studies focusing on the relationship between speciﬁc diagnoses and postoperative outcomes may fail to account for other psychological constructs that may be shared across diagnoses. Mood disorders, BED, and SUDs all share the common psychological construct of impulsivity, considered an important aspect of executive functioning. A lack of impulse control may contribute to the excessive weight gain seen in extreme obesity and may impact the results of bariatric surgery.

Disinhibition and Impulsivity among Persons with Extreme Obesity; Studies have suggested that individuals with obesity, and in particular those with extreme obesity presenting for bariatric surgery, show some deﬁcits in executive functioning. For example, candidates for bariatric surgery have shown deﬁcits in working memory, mental ﬂexibility, motor speed and complex attention.These deﬁcits could impact comprehension and retention of information presented to patients during the preoperative consultation process and, thus, negatively impact the ability to adhere to the dietary and behavioral changes required for an optimal postoperative outcome. At the same time, metabolic dysregulation, such as insulin resistance or hyperglycemeia seen in type 2 diabetes, also is associated with cognitive deﬁcits, suggesting a potential physiological mechanism for the relationship. Dietary disinhibition, deﬁned as a loss of control over eating, plays a central role in the overconsumption of food and, subsequently, the development of obesity. Disinhibition is similar to impulsivity, the term more commonly used in the substance use and smoking cessation literatures. Impulsivity is a multi-faceted construct and refers to the absence of the ability to inhibit an automatic behavior (otherwise known as response inhibition) and the tendency to discount future consequences in favor of more immediate outcomes (known as delay discounting). Similar to the role of disinhibition in obesity, impulsivity contributes to the development of and relapse with SUDs. Indeed, response inhibition and delay discounting are associated with both SUDs and obesity. Both also predict response to treatment for both SUDs and obesity. Chronic overeating and binge eating share several neurobiological and behavioral similarities with SUDs. In this regard, both may be viewed as behavioral disorders, in which intake (of food, alcohol, and/or drugs) escalates to a rate that is unhealthy and maladaptive. Nevertheless, the speciﬁc nature of the relationship between binge eating and substance use remains to be fully elucidated. There are similarities between binge eating and addictive disorders, including craving for the desired substance (drug or highly palatable food), a sense of loss of control when using, repeated attempts to control use despite clear adverse consequences, and the dedication of much time in obtaining and using the substance. Thus, the disinhibition observed with obesity and binge eating, the impulsivity seen with substance use disorders, and the emotional dysregulation associated with mood disorders all likely share commonalities that may both contribute to the development of extreme obesity and also may be associated with weight loss and changes in psychosocial status after bariatric surgery.

Psychosocial Status and Psychopathology after Bariatric Surgery:

In general, individuals who undergo bariatric surgery report dramatic improvements in psychosocial status and functioning postoperatively. The vast majority of patients report signiﬁcant reductions in symptoms of depression and anxiety in the ﬁrst postoperative year. They also report signiﬁcant improvements in health and weight-related quality of life. Patients also report improvements in body image, sexual functioning, and relationship satisfaction. The relationship between preoperative psychopathology and postoperative outcomes is less robust. Livhits and colleagues reviewed this literature and concluded that the preoperative factors of BMI, BED, and the presence of personality disorders provided the strongest negative associations with postoperative weight loss. At least two studies have suggested that preoperative psychopathology, particularly mood and anxiety disorders, is associated with smaller weight postoperative weight losses. The relationship between BED and postoperative weight loss is unclear; some studies have found a relationship between preoperative BED and postoperative weight loss while others have not. Additionally, two studies have suggested that a history of substance abuse is associated with larger weight losses following bariatric surgery. The interpretation of this counterintuitive ﬁnding is that the self-regulation skills that help patients maintain their sobriety also help patients adhere to the demands of the recommended postoperative diet.

Disinhibition and Impulsivity following Bariatric Surgery Encouragingly, studies have shown that there are improvements in executive functioning in persons with extreme obesity in the ﬁrst two years after bariatric surgery. Postoperatively, patients typically report decreases in disinhibition and hunger, as well as increases in cognitive restraint. The physical aspects of bariatric surgery typically prevent individuals from eating the objectively large amount of food necessary to meet the diagnostic criteria of BED. However, many individuals continue to report the feeling of loss of control over their eating.The self-reported inability to control these impulses postoperatively is associated with smaller weight losses and greater emotional distress in the ﬁrst few postoperative years. There is additional evidence that patients have difﬁculty with impulse control after surgery. A number of studies have suggested that there is an increased risk of substance abuse following bariatric surgery. King and colleagues, in their seminal investigation, found an increased rate of alcohol use disorder in the second postoperative year as compared to the year prior to surgery or in the ﬁrst postoperative year. Other recent studies also have found increases in alcohol or composite substance abuse (drug, alcohol, or cigarettes) in the ﬁrst two years after bariatric surgery. Postoperative substance use has been associated with smaller postoperative weight losses, postoperative nocturnal eating, and subjective hunger. Patients at greatest risk for new onset SUDs were more likely to report problems with high sugar/low fat food before surgery, further suggesting the role of impulsivity in eating behavior and substance use before and after surgery. This increase in substance abuse after surgery has been described as addiction transfer and characterized as a modern example of symptom substitution in which abuse of one substance (food) is replaced by another (alcohol or drugs) when patients are unable to consume large amounts of food after surgery. A potential contributor to addiction transfer may be emotional dysregulation. In general, symptoms of depression typically improve within the ﬁrst six months of bariatric surgery as patients are in the period of most rapid weight loss. Within the ﬁrst two postoperative years, the use of anti-depressant medications also decreases; however, a substantial minority of patients report using these medications two years after surgery. As most patients begin to regain weight postoperatively, they also experience an erosion of the improvements in depressive symptoms and quality of life. In addition, a higher-than-expected number of postoperative suicides have been documented. A secondary aim of the proposed study will investigate the relationship between changes in weight during the ﬁrst two postoperative years and changes in psychosocial status.

The proposed observational study will evaluate the relationship between measures of psychopathology, disordered eating, and impulsivity, (each assessed preoperatively and in the early postoperative period) and changes in weight and psychosocial status in the first two years after bariatric surgery. All participants will complete assessments at baseline (before surgery) and at 6, 12, and 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years old 18 years of age or above
* BMI of 35-60 kg/m2 (35 kg/m2 in the presence of signiﬁcant weight-related comorbidities, including established coronary artery disease, established peripheral arterial disease, symptomatic carotid artery disease, sleep apnea, metabolic syndrome, cardiomyopathy, hypertension, and debilitating joint pain).

Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure 160 or diastolic blood pressure 100mmHg)
* HbA1c 11%
* Recent history of cardiovascular disease (myocardial infarction or stroke within the past 6 months)
* Clinically signiﬁcant hepatic or renal disease Long-term treatment with oral steroids
* Current use of weight loss medication (OTC or prescription)
* Psychiatric hospitalization in the past 6 months
* Psychiatric diagnosis that would contraindicate surgery (e.g., schizophrenia)
* History of bariatric surgery
* Non-ambulatory individuals, deﬁned as those who are unable to walk without a cane or walker
* Lack of capacity to provide informed consent
* Plans to relocate from the area within 2 years
* Principal Investigator discretion

For the cognitive, computer-based testing:

* Any impairment (physical and/or neurological) including visual or other impairment preventing cognitive task performance
* Hearing impairment, significant hearing loss (more than 20% in either ear), cochlear implants, or bi-lateral hearing aids (will be assessed on a case-by-case basis to determine whether participants are eligible to complete the Stop Signal Task)
* Color Blindness (will be assessed on a case-by-case basis to determine whether participants are eligible to complete the Stroop Task)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Bariatric Surgery Programs at the Hospital of the University of Pennsylvania and Presbyterian Medical Center, all part of Penn Medicine. The investigators will enroll participants until a total of 300 adults have completed baseline visits. Based on the investigator's previous studies of bariatric surgery patients, the investigators expect that approximately 80% of participants will be women and 20% of participants will be ethnic minorities.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals interested in bariatric surgery attended an information session where the study was advertised. During a preoperative medical weight management visit with the program, the study was explained to patients. If they expressed interest, a brief screen was completed to assess eligibility. If patients met the inclusion criteria, they provided written informed consent to participate and were scheduled for study assessments. Recruitment occurred from 03/2016-11/2018.
Pre-assignment Details: We enrolled and assessed participants prior to bariatric surgery. Of the 300 enrolled, 281 underwent surgery, so 19 were not followed/contacted after the baseline assessment.
Groups:
- Patients Seeking Bariatric Surgery: We recruited 300 individuals seeking laparoscopic Roux-en-y gastric bypass or sleeve gastrectomy procedure and assessed them at baseline, 6, 12, and 24+ months following surgery.
Period: Overall Study
Arm/Group | Patients Seeking Bariatric Surgery
Started | 300
Completed | 227
Not Completed | 73

BASELINE CHARACTERISTICS:
Arm/Group | Patients Seeking Bariatric Surgery
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 224
  Unknown or Not Reported | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 179
  White | 87
  More than one race | 13
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change
Description: percent weight change from baseline
Time Frame: 6, 12, 24 months
Population: We had 245 participants at 6 months, 224 participants at 12 months, and 227 participants at 24 months complete a weight measurement that was available to compute percent weight change from baseline.
Measure: Mean (Standard Deviation); unit: percent weight change
Arm/Group | Patients Seeking Bariatric Surgery
Number analyzed (Participants) | 245
percent weight change
  % wt change at 6 mos | 23.0 (5.1)
  % wt change at 12 mos: number analyzed (Participants) | 224
  % wt change at 12 mos | 26.2 (7.7)
  % wt change at 24 mos: number analyzed (Participants) | 227
  % wt change at 24 mos | 23.3 (9.9)

ADVERSE EVENTS:
Time Frame: baseline (prior to surgery) through 24-36 months following surgery.
Description: Participants underwent bariatric surgery; we did not assess adverse events related to the surgery, only to completing the psychosocial assessment visits associated with the study.
Arm/Group | Patients Seeking Bariatric Surgery
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02775071/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT02775071/ICF_001.pdf